CLINICAL TRIAL: NCT01372774
Title: A Phase III Trial of Post-Surgical Stereotactic Radiosurgery (SRS) Compared With Whole Brain Radiotherapy (WBRT) for Resected Metastatic Brain Disease
Brief Title: Stereotactic Radiosurgery or Whole-Brain Radiation Therapy in Treating Patients With Brain Metastases That Have Been Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N107C; NCCTG-N107C; CDR0000701474 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-02676 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2011-06-11; First posted 2011-06-14 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Cognitive/Functional Effects; Metastatic Cancer; Neurotoxicity; Radiation Toxicity; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: neurotoxicity; radiation toxicity; cognitive/functional effects; tumors metastatic to brain; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neoplasm Metastasis; Neurotoxicity Syndromes; Radiation Injuries; Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I - WBRT (Active Comparator): Patients undergo whole brain radiotherapy (WBRT) once a day, 5 days a week, for approximately 3 weeks. Patient observation/follow up occurs at week 12 and months 6, 9, 12, 16 and 24 post registration/randomization. Event monitoring occurs every 6 months until 5 years post registration/randomization.
  Interventions: Radiation: whole-brain radiation therapy
- Arm II - SRS (Experimental): Patients undergo stereotactic radiosurgery (SRS) using a gamma knife or a linear accelerator procedure. Patient observation/follow up occurs at week 12 and months 6, 9, 12, 16 and 24 post registration/randomization. Event monitoring occurs every 6 months until 5 years post registration/randomization.
  Interventions: Radiation: stereotactic radiosurgery

INTERVENTIONS:
Radiation: stereotactic radiosurgery — Undergo RT
  Arms: Arm II - SRS
Radiation: whole-brain radiation therapy — Undergo radiotherapy (RT)
  Arms: Arm I - WBRT

SUMMARY:
RATIONALE: Stereotactic radiosurgery may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Radiation therapy uses high-energy x rays to kill tumor cells. It is not yet known whether stereotactic radiosurgery is more effective than whole-brain radiation therapy in treating patients with brain metastases that have been removed by surgery.

PURPOSE: This randomized phase III trial studies how well stereotactic radiosurgery works compared to whole-brain radiation therapy in treating patients with brain metastases that have been removed by surgery.

DETAILED DESCRIPTION:
Primary Goals

1. Overall Survival - To determine in patients with one to four brain metastases whether there is improved overall survival in patients who receive SRS to the surgical bed compared to patients who receive WBRT.
2. Neurocognitive Progression - To determine in patients with one to four brain metastases whether there is less neurocognitive progression post-randomization in patients who receive SRS to the surgical bed compared to patients who receive WBRT.

Secondary Goals

1. Quality of Life (QOL) - To determine in patients with resected brain metastases whether there is improved QOL in patients who receive SRS to the surgical bed compared to patients who receive WBRT.
2. Central Nervous System Failure - To determine in patients with one to four brain metastases whether there is equal or longer time to central nervous system (CNS) failure (brain) in patients who receive SRS to the surgical bed compared to patients who receive WBRT.
3. Functional Independence - To determine in patients with one to four brain metastases whether there is longer duration of functional independence in patients who receive SRS to the surgical bed compared to patients who receive WBRT.
4. Long-Term Neurocognitive Status - To determine in patients with one to four brain metastases whether there is better long-term neurocognitive status in patients who receive SRS to the surgical bed compared to patients who receive WBRT.
5. Adverse Events - To tabulate and descriptively compare the post-treatment adverse events associated with the interventions.
6. Local Tumor Bed Recurrence - To evaluate local tumor bed recurrence at 6 months with post-surgical SRS to the surgical bed in comparison to WBRT.
7. Local Recurrence - To evaluate time to local recurrence with post-surgical SRS to the surgical bed in comparison to WBRT.
8. CNS Failure Patterns - To evaluate if there is any difference in CNS failure patterns (local, distant, leptomeningeal) in patients who receive SRS to the surgical bed compared to patients who receive WBRT.

OUTLINE: This is a multicenter study. Patients are stratified according to age in years (< 60 vs ≥ 60), extracranial disease controlled (≤ 3 months vs > 3 months), number of pre-operative brain metastases (1 vs 2-4), histology (lung vs radioresistant [brain metastases from a sarcoma, melanoma, or renal cell carcinoma histology] vs other), and resection cavity maximal diameter (≤ 3 cm vs > 3 cm). Patient must complete baseline QOL and neurocognitive tests prior to registration/randomization. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo whole-brain radiotherapy (WBRT) once a day, 5 days a week, for approximately 3 weeks.
* Arm II: Patients undergo stereotactic radiosurgery (SRS) using a gamma knife or a linear accelerator procedure.

Event monitoring occurs up to 5 years post registration/randomization.

ELIGIBILITY:
Pre-registration Inclusion Criteria:

1. Number of Brain Metastases - Four or fewer brain metastases (as defined on the pre-operative MRI or CT brain scan) and status post resection of one of the lesions.
2. Non-CNS Primary Site - Pathology from the resected brain metastasis must be consistent with a non-central nervous system primary site. Note: Patients with or without active disease outside the nervous system are eligible (including patients with unknown primaries), as long as the pathology from the brain is consistent with a non-central nervous system primary site.
3. Size of Metastases - Any unresected lesions must measure < 3.0 cm in maximal extent on the contrasted MRI or CT brain scan obtained ≤ 35 days prior to pre-registration. The unresected lesions will be treated with SRS as outlined in the treatment section of the protocol. Note: The metastases size restriction does not apply to the resected brain metastasis; with resected brain metastases only surgical cavity size determines eligibility.
4. Size of Resection Cavity - Resection cavity must measure <5.0 cm in maximal extent on the post-operative MRI or CT brain scan obtained ≤35 days prior to pre-registration.

   Note: It is permissible for the resection of a dominant brain metastasis to include a smaller "satellite" metastasis as long as the single resection cavity is less than the maximum size requirements.
5. Tumor Staging Procedures - All standard tumor-staging procedures necessary to define baseline extra cranial disease status completed ≤42 days prior to pre-registration.
6. Treatment with Gamma Knife or Radiosurgery - Able to be treated with either a gamma knife or a linear accelerator-based radiosurgery system.
7. Age ≥ 18 years
8. Neurocognitive Testing - Willing and able to complete neurocognitive testing without assistance from family and companions. Note: Because neurocognitive testing is one of the primary goals of this study, patients must be able to utilize English language booklets (and/or French booklets if enrolled in Canada).
9. Quality of Life (QOL) Questionnaires - Willing and able to complete QOL by themselves or with assistance
10. ECOG Performance Status - ECOG Performance Status (PS) 0, 1, or 2.
11. SRS Credentialed by IROC Houston Quality Assurance - The site's SRS facility is IROC Houston Quality Assurance approved.
12. Neurocognitive Testing Credentialing - The site study team member performing neurocognitive testing of patients must have credentialing confirming completion of the neurocognitive testing training of the protocol.
13. Written Informed Consent - Provide written informed consent
14. Mandatory Samples for Correlative Tests - Willing to provide mandatory blood and urine samples for correlative research purposes.

Pre-registration Exclusion Criteria:

1. Pregnancy, Nursing and Contraception - pregnant women, nursing women and men or women of childbearing potential who are unwilling to employ adequate contraception throughout the study and for men for up to 3 months after completing treatment.
2. Prior Cranial Radiation Therapy
3. MRI or CT Scans - Inability to complete a MRI or CT scan with contrast of the head.
4. Gadolinium Allergy - Known allergy to gadolinium.
5. Cytotoxic Chemotherapy - Planned cytotoxic chemotherapy during the SRS or WBRT.
6. Other Tumor Types - Primary germ cell tumor, small cell carcinoma, or lymphoma
7. Leptomeningeal Metastasis - Widespread definitive leptomeningeal metastasis
8. Location of Brain Metastasis - A brain metastasis that is located ≤ 5 mm of the optic chiasm or within the brainstem.

Randomization Inclusion Criteria:

1. Number of Unresected Lesions - Post-operative MRI or CT scan confirmed zero, one, two or three unresected lesions.

   1.1 Each unresected lesion must measure ≤ 3.0 cm in maximal extent on the contrasted post-operative MRI or CT brain scan.

   1.2 Note: The pre-registration, post-operative, brain scan may be used for the randomization scan if obtained ≤ 28 days prior to randomization.

   1.3 Note: If there are no unresected brain metastases (i.e., all brain metastases have been resected), a post-operative CT brain scan may be used if obtained ≤ 28 days prior to randomization.
2. Size of Resection Cavity - Post-operative MRI or CT scan confirms resection cavity measures < 5.0 cm in maximal extent.

   2.1 Note: The pre-registration, post-operative brain scan may be used for the randomization scan if obtained ≤ 28 days prior to randomization.

   2.2 Note: If there are no unresected brain metastases (i.e., all brain metastases have been resected), a post-operative CT brain scan may be used if obtained ≤28 days prior to randomization.
3. Urine or Serum Pregnancy Test - Negative urine or serum pregnancy test done ≤ 7 days prior to randomization, for women of child bearing potential only.

Randomization Exclusion Criteria: none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2019-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul D. Brown, MD, Study Chair — M.D. Anderson Cancer Center
Locations (37):
- United States (37):
  - Mills - Peninsula Hospitals, Burlingame, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Mount Sinai Medical Center, Miami Beach, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Lowell General Hospital, Lowell, Massachusetts
  - Saint Vincent Hospital/Reliant Medical Group, Worcester, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sanford Clinic North-Bemidji, Bemidji, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Somerset Medical Center, Somerville, New Jersey
  - State University of New York Upstate Medical University, Syracuse, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Aria Health-Torresdale Campus, Philadelphia, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Huntoon K, Anderson SK, Ballman KV, Twohy E, Dooley K, Jiang W, An Y, Li J, von Roemeling C, Qie Y, Ross OA, Cerhan JH, Whitton AC, Greenspoon JN, Parney IF, Ashman JB, Bahary JP, Hadjipanayis C, Urbanic JJ, Farace E, Khuntia D, Laack NN, Brown PD, Roberge D, Kim BYS. Association of circulating markers with cognitive decline after radiation therapy for brain metastasis. Neuro Oncol. 2023 Jun 2;25(6):1123-1131. doi: 10.1093/neuonc/noac262. PMID 36472389
- [Derived] Palmer JD, Klamer BG, Ballman KV, Brown PD, Cerhan JH, Anderson SK, Carrero XW, Whitton AC, Greenspoon J, Parney IF, Laack NNI, Ashman JB, Bahary JP, Hadjipanayis CG, Urbanic JJ, Barker FG 2nd, Farace E, Khuntia D, Giannini C, Buckner JC, Galanis E, Roberge D. Association of Long-term Outcomes With Stereotactic Radiosurgery vs Whole-Brain Radiotherapy for Resected Brain Metastasis: A Secondary Analysis of The N107C/CEC.3 (Alliance for Clinical Trials in Oncology/Canadian Cancer Trials Group) Randomized Clinical Trial. JAMA Oncol. 2022 Dec 1;8(12):1809-1815. doi: 10.1001/jamaoncol.2022.5049. PMID 36264568
- [Derived] Brown PD, Ballman KV, Cerhan JH, Anderson SK, Carrero XW, Whitton AC, Greenspoon J, Parney IF, Laack NNI, Ashman JB, Bahary JP, Hadjipanayis CG, Urbanic JJ, Barker FG 2nd, Farace E, Khuntia D, Giannini C, Buckner JC, Galanis E, Roberge D. Postoperative stereotactic radiosurgery compared with whole brain radiotherapy for resected metastatic brain disease (NCCTG N107C/CEC.3): a multicentre, randomised, controlled, phase 3 trial. Lancet Oncol. 2017 Aug;18(8):1049-1060. doi: 10.1016/S1470-2045(17)30441-2. Epub 2017 Jul 4. PMID 28687377
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I - WBRT | Arm II - SRS
Started | 96 | 98
Completed | 92 | 93
Not Completed | 4 | 5
Not completed — Withdrawal prior to treatment | 4 | 5

BASELINE CHARACTERISTICS:
Population: All patients were included in baseline analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I - WBRT | Arm II - SRS | Total
Number analyzed (Participants) | 96 | 98 | 194
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [54 to 68] | 61 [54 to 66] | 61 [54 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 52 | 98
  Male | 50 | 46 | 96
Region of Enrollment [Number; unit: participants]
  North America | 96 | 98 | 194

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Deterioration Free Survival Post-radiation in Patients Who Received SRS Compared to Patients Who Received WBRT
Description: To determine in patients with one to four brain metastases whether there is less nuerocognitive progression post-randomization in patients who receive SRS to the surgical bed compared to patients who receive WBRT. Neurocognitive progression is defined as a drop of at least one stanard deviation from baseline in one of the six neurocognitive tests at post-randomization evaluation.
Time Frame: from baseline up to 5 years post radiation
Population: All enrolled patients were included in the analysis of this outcome. This includes the 9 patients that did not receive treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I - WBRT | Arm II - SRS
Number analyzed (Participants) | 96 | 98
Months | 3.0 [2.86 to 3.25] | 3.7 [3.45 to 5.06]
Statistical Analysis 1: Comparison: Arm I - WBRT vs Arm II - SRS; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.35 to 0.63]

2. Primary Outcome: Overall Survival
Description: To determine in patients with one to four brain metastases whether there is improved overall survival in patients who receive SRS to the surgical bed compared to patients who receive WBRT. Overall survival is defined as the time from randomization to death from any cause.
Time Frame: from baseline up to 5 years post radiation
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I - WBRT | Arm II - SRS
Number analyzed (Participants) | 96 | 98
months | 11.6 [9.9 to 18] | 12.2 [9.7 to 16.3]
Statistical Analysis 1: Comparison: Arm I - WBRT vs Arm II - SRS; Test type: Superiority; p = 0.70, Log Rank; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.76 to 1.50]

3. Secondary Outcome: Local Control of the Surgical Bed
Description: Local control of the surgical bed means that tumor did not recur at the unresected metastases treated with stereotactic radiosurgery, SRS, or whole brain radiotherapy, WBRT. Intercranial Brain Control Rates estimated via 1-Cumulatice Incidence Rate from Competing Risk survival analysis of time to the specific recurrence type. Deaths without recurrence are censored at time of death.
Time Frame: Up to 6 months post radiation
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm I - WBRT | Arm II - SRS
Number analyzed (Participants) | 96 | 98
percentage of patients | 87.1 [80.5 to 94.2] | 80.4 [72.8 to 88.7]
Statistical Analysis 1: Comparison: Arm I - WBRT vs Arm II - SRS; Test type: Superiority; p = 0.00068, Gray's K-sample — Intracranial Brain Control Rates estimated via 1-Cumulative Incidence Rate from Competing Risk survival analysis of time to the specific recurrence type. Deaths without recurrence are censored at time of death

4. Secondary Outcome: Time to CNS Failure in These Patients
Time Frame: Up to 5 years post radiation
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I - WBRT | Arm II - SRS
Number analyzed (Participants) | 96 | 98
Months | 27.5 [14.85 to NA] — Not Reached | 6.4 [5.16 to 8.90]

5. Secondary Outcome: Change in Quality-of-life at 6 Months
Description: Clinically significant change in quality of life is defined as ten-point change on QOL scores (transformed to a 0 to 100 scale). As measured by the overall score from the FACT-Br. An improvement is defined as a change greater than or equal ten points.
Time Frame: Up to 6 months post randomization
Population: Only patients with baseline and 6 month QOL assessment scores were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Arm I - WBRT | Arm II - SRS
Number analyzed (Participants) | 64 | 65
participants
  Improvement | 4 | 6
  Stable | 24 | 33
  Decline | 17 | 12
  Missing | 19 | 14
Statistical Analysis 1: Comparison: Arm I - WBRT vs Arm II - SRS; Test type: Superiority; p = 0.31, Chi-squared

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: CTCAE term (AE description) and grade: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. All appropriate treatment areas should have access to a copy of the CTCAE version 4.0. A copy of the CTCAE version 4.0 can be downloaded from the CTEP website (http://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm)
Arm/Group | Arm I - WBRT | Arm II - SRS
Serious Adverse Events (participants affected / at risk) | 14/92 | 19/93
Other Adverse Events (participants affected / at risk) | 74/92 | 64/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - WBRT (N=92) | Arm II - SRS (N=93)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Optic nerve disorder (Eye disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 0 (0)
Death NOS (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Sudden death NOS (General disorders) | 1 (1) | 0 (0)
Esophageal infection (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pancreas infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Hemoglobin increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Central nervous system necrosis (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (3) | 2 (4)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Thromboembolic event (Vascular disorders) | 1 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - WBRT (N=92) | Arm II - SRS (N=93)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 1 (2)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 6 (12) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 21 (62) | 15 (46)
Middle ear inflammation (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 2 (5) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1)
Optic nerve disorder (Eye disorders) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 4 (7)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 36 (65) | 22 (31)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 21 (24) | 9 (13)
Death NOS (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 20 (31) | 10 (23)
Gait disturbance (General disorders) | 1 (2) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 14 (19) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (3) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Weight gain (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 2 (5) | 1 (2)
White blood cell decreased (Investigations) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (8) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (7) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 0 (0) | 6 (8)
Cognitive disturbance (Nervous system disorders) | 27 (52) | 17 (26)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 4 (5)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 3 (3) | 0 (0)
Meningismus (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 10 (16) | 16 (23)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 3 (3) | 6 (6)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Uterine hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 49 (119) | 28 (57)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No